CLINICAL TRIAL: NCT06720129
Title: The Application Effect of Modified Pressure-Reducing Fixation Protective Nasal Strip in the Nursing Care of Patients Receiving High-Flow Nasal Cannula Therapy
Acronym: HFNC; pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ying Zhou (Other Government)
Responsible Party: Sponsor-Investigator, Ying Zhou, Principal Investigator, Wuxi Ninth People's Hospital
Organization: Wuxi Ninth People's Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: KS2024035
Record Dates: First submitted 2024-11-21; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: High-Flow Nasal Cannula Therapy
Keywords: HFNC; pressure ulcer; patient comfort; Modified Pressure-Reducing Fixation Protective Nasal Strip; nursing efficacy
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group (Other): The control group received standard care plus a hydrocolloid dressing for protection
  Interventions: Device: Standard care alone
- The observation group (Other): The observation group employed the modified pressure-reducing fixation protective nasal strip
  Interventions: Device: the modified pressure-reducing fixation protective nasal strip

INTERVENTIONS:
Device: the modified pressure-reducing fixation protective nasal strip — Materials Preparation consists of one foam dressing, one piece of 3M tape, and two pairs of scissors. 2. Manufacturing Procedure: step 1 Cut the foam dressing into two large rectangles and one little T-shape based on the patient's face shape and size as well as the width of the nasolabial fold. Attach these sections to the nasolabial fold region and both cheeks, respectively . Step 2: Based on the size of the oxygen cannula, set up small, medium, and large fixation patch models. Select the appropriate model according to the patient's condition and make the necessary cuts to properly secure the nasal prongs. Step 3: Check the tightness of the head strap, ensuring it is snug enough to fit one finger beneath it to avoid pressing on the skin around the ears. Ensure proper placement on the patient. See Figure 1 for detailed application.
  Arms: The observation group
Device: Standard care alone — standard care plus a hydrocolloid dressing for protection
  Arms: The control group

SUMMARY:
This study was a prospective, randomized controlled trial that included 60 patients receiving high-flow nasal cannula (HFNC) therapy. Participants were randomly divided into two groups: the observation group (n=30), which used a modified decompression fixation protective patch, and the control group (n=30), which received hydrocolloid dressing protection in addition to standard care. The study compared general demographic data, the interval time between changing fixation straps, the times of adjusting the catheter position, the effectiveness of skin management, the number of ineffective oxygenation attempts, the incidence of adverse events, and patient comfort scores between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* 1. Meet the diagnostic criteria for respiratory failure, worsening dyspnea, acute exacerbation of chronic obstructive pulmonary disease (COPD), bronchitis, pneumonia, and congestive heart failure.
* 2. No severe cognitive impairment.
* 3. Good compliance and being able to actively cooperate with the investigation.
* 4. No concurrent metabolic diseases.

Exclusion Criteria:

* 1. Patients with severe respiratory failure, severe arrhythmias, concurrent pneumothorax, coma upon admission, or persistent vomiting.
* 2. Patients with severe liver failure, kidney failure, or other severe systemic diseases.
* 3. Patients with severe cognitive impairment who are unable to understand or comply with the study requirements.
* 4. Patients with severe hemodynamic instability.
* 5. Patients with allergies to oxygen therapy or protective patch materials.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Interval Time for Changing the Fixation Strap | The time from receiving high-flow nasal cannula (HFNC) therapy to removal as per medical advice. up to a month.
Times of Adjusting the Catheter Position | Data were collected every three days from the initiation of high-flow nasal cannula (HFNC) therapy until its removal as per medical advice. up to a month.
Effectiveness of skin management | The time from receiving high-flow nasal cannula (HFNC) therapy to removal as per medical advice. up to a month.
  The Braden Scale assesses six factors to determine a patient's risk of developing pressure ulcers. Each factor is scored from 1 to 4 (except for activity and friction/shear, which are scored from 1 to 3), with a total possible score of 23. The lower the total score, the higher the risk of pressure ulcers. (Sensory Perception: Assesses the patient's ability to perceive and respond to discomfort or pressure on the skin; Normal sensation: 4 points. Completely unable to sense: 1 point. Moisture: Evaluates the frequency of skin exposure to moisture. Skin stays dry: 4 points; Skin is often moist: 1 point. Activity: Assesses the patient's ability to move. Fully mobile: 4 points; Completely bedridden: 1 point. Mobility: Evaluates the patient's ability to change and control body position. Fully able to move and control: 4 points; Completely unable to move: 1 point. Nutrition: Assesses the patient's nutritional intake. Good nutrition: 4 points; Very poor nutrition: 1 point. Friction and Shear:
Incidence of Ineffective Oxygenation | The time from receiving high-flow nasal cannula (HFNC) therapy to removal as per medical advice. up to a month.

SECONDARY OUTCOMES:
Comparison of Comfort Levels | Assessed on the 3th day after the start of the experiment
  Patient comfort is assessed on the 3th day after the start of the experiment. The scale includes 4 dimensions with 30 items, scored from 30 to 120. Higher scores indicate greater comfort. Total score < 60: Low comfort; Score 60-90: Moderate comfort; Score > 90: High comfort.
Adverse Event Incidence | The time from receiving high-flow nasal cannula (HFNC) therapy to removal as per medical advice. up to a month.
  adverse events such as nasal mucosal indentation, nasal mucosal pain, nasal pressure injuries, catheter dislodgement, and medical adhesive-related skin injuries.

OTHER OUTCOMES:
Gender | The time from admission to discharge. up to 6 weeks.
Age | The time from admission to discharge. up to 6 weeks.
Length of hospital stay | The time from admission to discharge. up to 6 weeks.
Days of treatment use | The time from admission to discharge. up to 6 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuxi Ninth People's Hospital, Wuxi, Jiangsu, China